CLINICAL TRIAL: NCT00005378
Title: Impact of Sleep Disordered Breathing in Older Adults
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4276; R01HL051075 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2001-11

CONDITIONS: Cardiovascular Diseases; Hypertension; Depression; Sleep Apnea Syndromes; Lung Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Depression; Sleep Apnea Syndromes; Lung Diseases

SUMMARY:
To test the hypothesis that clinically inapparent sleep-disordered breathing was associated with blood pressure elevation, impairment of health-related quality of life, and depression.

DETAILED DESCRIPTION:
BACKGROUND:

The health impact of disordered breathing during sleep among middle-aged and older men and women in the general population had not been well studied, and the need for treating relatively mild degrees of sleep-disordered breathing was unknown in 1994. The study was the first population study which examined the effect of sleep-disordered breathing on these health outcomes. The study sought to establish the prevalence of clinically important sleep-disordered breathing among middle-aged and older men and women and to provide quantitative data to serve as the basis for selecting patients for screening and deciding which patients might benefit from therapeutic intervention.

DESIGN NARRATIVE:

The study evaluated the hypothesis that clinically inapparent sleep-disordered breathing was associated with blood pressure elevation, impairment of health-related quality of life, and depression. The study used the Veterans Administration Normative Aging Study (NAS) population, which consisted of approximately 1,700 community-dwelling-men who returned for examination every three years. Respiratory function was assessed during sleep among these men and their wives using a validated method for home sleep monitoring. Blood pressure, health-related quality of life, and depression score were also assessed in the home. The potential associations of sleep-disordered breathing with hypertension, impaired health-related quality of life, and depression were evaluated, and the possibility that these relationships differed between men and women was examined.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-07; Study Completion 1998-05 (Actual)